CLINICAL TRIAL: NCT02690506
Title: The Effect of Pregabalin on the Spinal Anesthesia: Randomized Controlled Placebo Study
Brief Title: The Effect of Pregabalin on the Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2014-05-027
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Block
Keywords: pregabalin; spinal anesthesia
MeSH Terms: conditions — Bites and Stings | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Group C (Placebo Comparator): Oral placebo pill was administered 2 hours before anesthesia
  Interventions: Drug: Placebo
- Group P (Active Comparator): Oral pregabalin 150 mg was administered 2 hours before anesthesia
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Placebo
  Arms: Group C
Drug: Pregabalin
  Arms: Group P

SUMMARY:
Pregabalin, an anticonvulsant is widely used for treatment of neuropathic pain. Recently, it was reported that premedication of pregabalin before general anesthesia is effective to reduce postoperative pain. Up to date, there is no study about the effect of premedication of pregabalin on the spinal anesthesia. Therefore, in this study, investigators investigate the effect of premedication of pregabalin on the spinal anesthesia.

DETAILED DESCRIPTION:
In this study, investigators investigate the effect of premedication of pregabaline 150 mg on the spinal anesthesia. Two hours before spinal anesthesia, placebo pill was administered to patients in the group C and pregabalin 150 mg was administered to patients in the group P, respectively. Time for the onset of blockade, cephalad level of analgesia and duration of analgesia were measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anaesthesiologists Grades I and II

Exclusion Criteria:

* Patients with infection at the puncture site, coagulopathy, having true hypersensitivity to drugs used, diabetes and hypertension, psychiatric and neurological diseases

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Duration of spinal anesthesia | 24 hours after spinal anesthesia
  Duration of spinal anesthesia was measured 24 after spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Dr, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea